CLINICAL TRIAL: NCT01282814
Title: Randomized, 2-way Crossover, Bioequivalence Study of Venlafaxine Hydrochloride 150 mg Extended-Release Capsules and Effexor® XR 150 mg Extended-Release Capsules Administered as the Content of 1 x 150 mg Extended-Release Capsule Mixed With Applesauce in Healthy Subjects Under Fasting Conditions.
Brief Title: Venlafaxine Hydrochloride 150 mg Extended-Release Capsules Sprinkle Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals, USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 30024
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Venlafaxine Hydrochloride

ARMS (2):
- Investigational Test Product (Experimental): Venlafaxine Hydrochloride 150 mg Extended-Release Capsules.
  Interventions: Drug: Venlafaxine Hydrochloride
- Reference Listed Drug (Active Comparator): Effexor® XR 150 mg Extended-Release Capsules
  Interventions: Drug: Effexor® XR

INTERVENTIONS:
Drug: Venlafaxine Hydrochloride — 150 mg Extended-Release Capsule
  Arms: Investigational Test Product
Drug: Effexor® XR — 150 mg Extended-Release Capsule
  Other Names: Venlafaxine Hydrochloride (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of venlafaxine hydrochloride 150 mg capsules (test) versus Effexor® XR (reference) administered as the content of 1 x 150 mg extended-release capsule mixed with applesauce under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Members of the community at large.
* Subjects will be females and/or males, non-smokers, 18 years of age and older.
* Female subjects will be postmenopausal or surgically sterilized.

Exclusion Criteria:

* Clinically significant illness within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities at screening.
* Subjects with BMI greater than 30.0.
* History of significant alcohol abuse within 6 months of the screening visit or any indication of the regular use of more than 14 units of alcohol per week (1 unit is equal to 150 mL of wine, 360mL of beer, or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, PCP, crack) within 1 year of the screening visit.
* History of allergic reactions to venlafaxine.
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* History or presence of any clinically significant gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products within 7 days prior to administration of study medication, except for topical products without systemic exposure.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Any food allergies, intolerance, restriction, or special diet that, in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* Subjects who have had a depot injection or implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:

  * less than 300 mL of whole blood within 30 days or
  * 300 mL to 500 mL of whole blood within 45 days or
  * more than 500 mL of whole blood within 56 days.
* Subjects who have consumed food or beverages containing grapefruit within 7 days prior to administration of the study medication.
* Subjects with clinically significant presence or history of raised intra-ocular pressure or at the risk of acute narrow angle glaucoma.
* Subjects who have dentures or braces.
* Intolerance to venipunctures.
* Subjects with a clinically significant history of tuberculosis, epilepsy, asthma, diabetes, or psychosis will not be eligible for this study.
* Subjects who are unable to understand or unwilling to sign the Informed Consent Form.
* Subjects with the known presence of volume-depletion.
* Subjects predisposed to bleeding of the skin and mucous membrane (impaired platelet aggregation).
* Subjects with clinically significant history of seizures.
* Additional exclusion criteria for females only:

  * Breastfeeding subjects.
  * Positive urine pregnancy test screen at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-02; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Venlafaxine Hydrochloride (Test) First: 150 mg Venlafaxine Hydrochloride Extended-Release Capsules test product dosed in first period followed by 150 mg Effexor® XR Capsules reference product dosed in the second period.
- Effexor® XR (Reference) First: 150 mg Effexor® XR Extended-Release Capsules reference product dosed in first period followed by 150 mg Venlafaxine Hydrochloride Extended-Release Capsules test product dosed in the second period.
Period: First Intervention
Arm/Group | Venlafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Started | 12 | 12
Completed | 12 | 9
Not Completed | 0 | 3
Not completed — Emesis During Dosing Interval | 0 | 3
Period: Washout of 7 Days
Arm/Group | Venlafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Started | 12 | 9
Completed | 10 | 9
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention
Arm/Group | Venlafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Caucasian | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Venlafaxine.
Description: Bioequivalence based on Venlafaxine Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Venlafaxine Hydrochloride (Test): 150 mg Venlafaxine Hydrochloride Extended-Release Capsules test product dosed in either period.
- Effexor® XR (Reference): 150 mg Effexor® XR Extended-Release Capsules reference product dosed in either period.
Arm/Group | Venlafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 19 | 19
ng/mL | 120.07 (45.48) | 103.59 (39.47)
Statistical Analysis 1: Comparison: Venlafaxine Hydrochloride (Test) vs Effexor® XR (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 115.85, 90% CI 2-sided [108.45 to 123.72] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Venlafaxine.
Description: Bioequivalence based on Venlafaxine AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Venlafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 1972.77 (1425.56) | 1800.03 (1270.77)
Statistical Analysis 1: Comparison: Venlafaxine Hydrochloride (Test) vs Effexor® XR (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 109.97, 90% CI 2-sided [103.68 to 116.63] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Venlafaxine.
Description: Bioequivalence based on Venlafaxine AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Venlafaxine Hydrochloride (Test) | Effexor® XR (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 2163.77 (1647.47) | 2065.50 (1626.52)
Statistical Analysis 1: Comparison: Venlafaxine Hydrochloride (Test) vs Effexor® XR (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 106.46, 90% CI 2-sided [101.45 to 111.71] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 2 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Venlafaxine Hydrochloride (Test) First | Effexor® XR (Reference) First
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 16/24 | 9/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venlafaxine Hydrochloride (Test) First (N=24) | Effexor® XR (Reference) First (N=24)
Tachycardia (General disorders) | 3 (4) | 0 (0)
Nausea (General disorders) | 7 (8) | 6 (8)
Jaw Stiffness (General disorders) | 2 (2) | 0 (0)
High Blood Pressure (General disorders) | 4 (4) | 0 (0)
Headache (General disorders) | 0 (0) | 2 (2)
Drowsiness (General disorders) | 0 (0) | 2 (2)
Loose Stools (General disorders) | 2 (2) | 2 (2)
Dizziness (General disorders) | 3 (4) | 1 (1)
Bradycardia (General disorders) | 2 (2) | 0 (0)
Vomiting (General disorders) | 0 (0) | 4 (4)
Hot Flushes (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.